CLINICAL TRIAL: NCT05010824
Title: Effects of Parent-based Educational Programme for Sleep Problems in Children With Autism Spectrum Disorder (ASD): A Randomized Controlled Trial
Brief Title: A Brief Parent-based Sleep Intervention for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW20-204
Record Dates: First submitted 2021-08-05; First posted 2021-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: ASD; Insomnia
Keywords: Sleep; ASD; Insomnia; Behavioral Intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention will involve three consultation sessions and four follow-up phone calls with parents to help them learn sleep hygiene practices and specific behavioural strategies to improve their child's sleep and follow up on the progress.
  Interventions: Behavioral: Sleep hygiene practices and behavioural intervention
- Waiting-list control (No Intervention): Children in the waiting-list control group will receive usual clinical care.

INTERVENTIONS:
Behavioral: Sleep hygiene practices and behavioural intervention — The first session will involve the provision of sleep-related psycho-education (e.g. sleep hygiene practices) and specific strategies to tackle problematic sleep-related behaviours, as well as collaborative goal setting and development of management plan tailored to the child's sleep problem. The second and third session will involve a review of the sleep diary and a reinforcement of learned strategies, and focus on problem-solving to tackle any issues that have emerged from implementing the behavioural strategies at home. Follow-up phone calls provide parents with an opportunity to ask any further questions and to consolidate learned strategies and further troubleshoot.
  Arms: Intervention group

SUMMARY:
Sleep problems are very common in children with ASD, with a prevalence rate as high as 78%, and often pose significant challenges and stress to the families. Sleep problems in children with ASD are strongly associated with the exacerbation of daytime symptoms, and poor parental sleep quality and mental health. The present study is a randomised controlled trial to compare the effects of a parent-based sleep intervention for children with ASD (aged 3-6). Eligible participants will be randomised to either intervention (three consultation sessions and four follow-up phone calls) or waiting-list control condition. Assessments will be conducted at pre-treatment (baseline), and one-week after the intervention (post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers (aged 21 or above) of preschool children (aged 3 to 6 years old) with a clinical diagnosis of ASD attending paediatric developmental clinic or clinical psychology service at the Duchess of Kent Child Assessment Centre (DKCAC)
* Clinical diagnosis of ASD would be made by either a Pediatrician or a Clinical Psychologist, using at least one of the following diagnostic tools: Childhood Autism Rating Scale, Second Edition (CARS-2), Autism Diagnostic Observation Schedule, Second Edition (ADOS-2), Autism Diagnostic Interview-Revised (ADI-R) and clinical interview based on diagnostic criteria of ASD depicted in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

Exclusion Criteria:

- Parent/caregiver of children with diagnosed co-morbid neurological, psychiatric or medical conditions which could have affected their sleep, such as obstructive sleep apnea, epilepsy, childhood anxiety disorder

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Child: Change of child's sleep | Baseline, immediately after the treatment
  Change of the child's sleep measured by the Children's Sleep Habits Questionnaire (CSHQ). The total score of CSHQ ranges from 33 to 99. A higher score reflects more sleep disturbance.
Child: change of insomnia symptoms (bedtime resistance) | Baseline, immediately after the treatment
  Change of the child's bedtime resistance measured by the Children's Sleep Habits Questionnaire (CSHQ) bedtime resistance score (6 items; score range: 6-18)
Child: change of insomnia symptoms (sleep onset delay) | Baseline, immediately after the treatment
  Change of the child's sleep onset delay measured by the Children's Sleep Habits Questionnaire (CSHQ) sleep onset delay score (1 item; score range: 1-3)
Child: change of insomnia symptoms (night waking) | Baseline, immediately after the treatment
  Change of the child's night waking measured by the Children's Sleep Habits Questionnaire (CSHQ) night waking score (3 items; score range: 3-9)

SECONDARY OUTCOMES:
Parent: Change of parental self-reported sleep quality | Baseline, immediately after the treatment
  Pittsburgh Sleep Quality Index (PSQI), a validated 19-item measure used to assess sleep habits, quality, and quantity, producing a total score and seven sub-scores in sleep quality, sleep onset latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The global score can range from 0 to 21. Higher scores suggest poorer sleep quality.
Parent: Change of parental insomnia symptoms | Baseline, immediately after the treatment
  Insomnia Severity Index (ISI). Total score ranges from 0-28 and higher scores indicate greater insomnia severity.
Child: Change of child's behaviour & other clinical symptoms | Baseline, immediately after the treatment
  Strengths and Difficulties Questionnaire - parent report, which is a 25-item screening measure for emotional and behavioral problems in children. It consists of five subscales. Each of the subscales consists of five items, and scale scores range from 0-10. A higher score is indicative of more problems for all subscales, except for the prosocial scale, where higher scores correspond to fewer difficulties in prosocial behaviour.
Child: Change of child's executive functions reported by parents | Baseline, immediately after the treatment
  Behavioral Rating Inventory of Executive Function - Preschool Version (BRIEF-P). It consists of 63 items that measure various behavioral manifestations of EF based on parent or teacher ratings, within the context of the child's everyday environment.
Parent: Change of parental mood symptoms | Baseline, immediately after the treatment
  Depression Anxiety Stress Scales - 21 item (DASS-21) consists of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items. Higher scores suggest more depression, anxiety and stress, respectively.
Parent: Change of parental stress | Baseline, immediately after the treatment
  Chinese version of Parental Stress Scale (PSS). It contains 17 items representing pleasure or positive themes of parenthood (emotional benefits, self-enrichment, personal development) and negative components (demands on resources, opportunity costs and restrictions). Higher scores on the scale indicate greater stress.
Parent: Change of parental sense of competence and satisfactory in parenting | Baseline, immediately after the treatment
  Parental Sense of Competence Scale (PSOC), which is a scale designed to measures parental competence on two dimensions: Satisfaction and Efficacy. It is a 16-item Likert-scale questionnaire (on a 6-point scale ranging from strongly agree [1] to strongly disagree [6]), with nine questions under Satisfaction and seven under Efficacy.
Parent: Parent's satisfaction to the treatment | Baseline, immediately after the treatment
  Treatment satisfaction rating scale, a parent-report measure specifically designed for the study. Lower scores suggest higher parental satisfaction.
Parent: Parent's overall health status | Baseline, immediately after the treatment
  Short Form 12-item Health Survey (SF-12v2), a validated measure of health-related quality of life (HRQOL). It consists of 12 items that cover 8 subscales, namely physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH). The eight subscale scores can be aggregated into a physical component summary (PCS) score and a mental component summary (MCS) score. Each of the eight SF-12v2 subscale has a scoring range from 0 to 100; a higher score indicates better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD,DClinPsy, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Clinical Psychology, The Duchess of Kent Children's Hospital at Sandy Bay, HKWC, Hospital Authority, Hong Kong
  - Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05010824/Prot_000.pdf